CLINICAL TRIAL: NCT00993187
Title: A Multicenter, Randomized, Double Blind Study to Compare the Efficacy and Safety of Sitagliptin/Metformin Fixed-Dose Combination (Janumet®) Compared to Glimepiride in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Sitagliptin/Metformin Fixed-Dose Combination (FDC) Compared to Glimepiride in Participants With Type 2 Diabetes Mellitus (MK-0431A-202)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431A-202; 2009_672 (Other: Merck Registration Number)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin/Metformin FDC (Experimental): Participants in the Sitagliptin/Metformin Fixed- Dose Combination (Sita/Met FDC) group received tablets of Sita/Met FDC and placebo tablets matching glimepiride for 30 weeks. The dose for Sita/Met FDC was 50/500 mg twice daily (b.i.d.) starting Day 1 and increased to 50/1000 mg b.i.d. over a period of 4 weeks.
  Interventions: Drug: Sitagliptin/Metformin FDC; Drug: Matching placebo to glimepiride
- Glimepiride (Active Comparator): Participants in the Glimepiride group received 2 placebo tablets matching Sita/Met FDC and glimepiride tablets (1 mg or 2 mg) for 30 weeks. The dose for glimepiride was 1 mg once daily (q.d.) starting Day 1 and up-titrated as considered appropriate by the investigator based upon the results of participant's self-monitored blood glucose levels but not to exceed 6 mg/day.
  Interventions: Drug: Comparator: Glimepiride; Drug: Matching placebo to Sitagliptin/Metformin FDC

INTERVENTIONS:
Drug: Sitagliptin/Metformin FDC — Sitagliptin phosphate plus metformin hydrochloride combination tablet (MK-0431A) orally up to 50/1000 mg BID for 30 weeks
  Other Names: Janumet®
  Arms: Sitagliptin/Metformin FDC
Drug: Comparator: Glimepiride — Glimepiride tablet orally up to 6 mg daily for 30 Weeks
  Other Names: Amaryl®
  Arms: Glimepiride
Drug: Matching placebo to Sitagliptin/Metformin FDC — Matching placebo to Sitagliptin/Metformin FDC 50/1000 mg orally BID for 30 weeks
  Arms: Glimepiride
Drug: Matching placebo to glimepiride — Matching placebo to glimepiride tablet orally daily for 30 weeks
  Arms: Sitagliptin/Metformin FDC

SUMMARY:
This study will assess the effect of sitagliptin/metformin FDC 50/1000 mg (Janumet®), MK-0431A) compared with the effect of glimepiride on hemoglobin A1c (HbA1c). The primary hypothesis is that after 30 weeks, sitagliptin/metformin FDC 50/1000 mg provides superior reduction in HbA1c (mean change from baseline) compared to glimepiride.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus
* Is currently not on an anti-hypoglycemic agent (AHA) (off for at least 12 weeks) and has a Visit 1/Screening Visit HbA1c greater than or equal to 7.0% and less than or equal to 9.5%; or is currently on AHA monotherapy or low-dose oral combination therapy (i.e., less than or equal to 50% maximum labeled dose of each agent) and has a Visit 1/Screening Visit HbA1c greater than or equal to 6.5% and less than or equal to 9.0%

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus or a history of ketoacidosis
* Has been on any investigational or approved glucagon-like peptide-1 (GLP-1) analogue (such as exenatide, liraglutide, etc.), any investigational or approved dipeptidyl peptidase IV (DPP-4) inhibitor (such as sitagliptin, vildagliptin, alogliptin, etc.) or a peroxisome proliferator-activated receptor (PPAR) gamma agonist agent (such as rosiglitazone, pioglitazone, etc.) within 12 weeks of Visit 1
* Required insulin within the prior 12 weeks
* Has a hypersensitivity or contraindication to any sulfonylurea medication (such as glimepiride, glipizide, etc.), DPP-4 inhibitor (such as sitagliptin, vildagliptin, alogliptin, etc.), or biguanide medication (such as metformin, etc.)
* Has inadequately controlled hypertension
* Has cirrhosis or active liver disease
* Has severe cardiac conditions
* Is obese
* Has human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2010-05-04 (Actual); Primary Completion 2013-10-29 (Actual); Study Completion 2013-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kim SS, Kim IJ, Lee KJ, Park JH, Kim YI, Lee YS, Chung SC, Lee SJ. Efficacy and safety of sitagliptin/metformin fixed-dose combination compared with glimepiride in patients with type 2 diabetes: A multicenter randomized double-blind study. J Diabetes. 2017 Apr;9(4):412-422. doi: 10.1111/1753-0407.12432. Epub 2016 Aug 8. PMID 27229178
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0431A-202&kw=NCT00993187&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Sitagliptin/Metformin: Participants in the Sitagliptin/Metformin Fixed- Dose Combination (Sita/Met FDC) group received tablets of Sita/Met FDC and placebo tablets matching glimepiride for 30 weeks. The dose for Sita/Met FDC was 50/500 mg twice daily (b.i.d.) starting Day 1 and increased to 50/1000 mg b.i.d. over a period of 4 weeks.
Period: Overall Study
Arm/Group | Sitagliptin/Metformin | Glimepiride
Started | 147 | 145
Received at Least 1 Dose of Study Drug | 146 | 144
Completed | 121 | 108
Not Completed | 26 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Metformin | Glimepiride | Total
Number analyzed (Participants) | 147 | 145 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.8 (8.5) | 53.1 (9.2) | 53.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 61 | 127
  Male | 81 | 84 | 165

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1C (HbA1C) at Week 30
Description: HbA1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%). Change in A1C following 30 weeks of therapy (i.e., A1C at Week 30 minus A1C at baseline).
Time Frame: Baseline and Week 30
Population: Full-Analysis-Set (FAS) Population included all randomized participants who had a baseline measurement, consumed at least one dose of study medication, and had at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of total hemoglobin
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 138 | 137
Percent of total hemoglobin | -1.5 [-1.6 to -1.4] | -0.7 [-0.8 to -0.6]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -0.8, 95% CI 2-sided [-1.0 to -0.6]

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 32 weeks
Population: The All Patients as Treated (APaT) Population includes all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 146 | 144
Participants | 88 | 101

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the product.
Time Frame: Up to 30 weeks
Population: The APaT Population includes all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 146 | 144
Participants | 8 | 8

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 30
Description: Blood glucose was measured on a fasting basis (collected after an 8- to 10-hour fast). FPG is expressed as mg/dL. Blood was drawn at predose on Day 1 and after 30 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 30 minus FPG at baseline).
Time Frame: Baseline and Week 30
Population: The FAS Population included all randomized participants who had a baseline measurement, consumed at least one dose of study medication, and had at least one post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 138 | 137
mg/dL | -47.0 [-51.7 to -42.3] | -23.5 [-28.2 to -18.8]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -23.5, 95% CI 2-sided [-30.0 to -16.9]

5. Secondary Outcome: Percentage of Participants With One or More Episodes of Hypoglycemia
Description: Symptomatic episodes assessed as likely to be due to hypoglycemia were reported by investigators as adverse experiences of hypoglycemia. Adverse experiences of hypoglycemia were based on all reports of hypoglycemia; a concurrent glucose measurement was not required.
Time Frame: Up to Week 30
Population: The APaT Population includes all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 146 | 144
Percentage of participants | 5.5 | 20.1
Statistical Analysis 1: Comparison: Sitagliptin/Metformin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in percent = -14.7, 95% CI 2-sided [-23.0 to -7.0]

6. Secondary Outcome: Change From Baseline in Body Weight at Week 30
Description: Change in body weight following 30 weeks of therapy (i.e., body weight at Week 30 minus body weight at baseline)
Time Frame: Baseline and Week 30
Population: The APaT Population includes all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 146 | 144
kg | -0.83 (1.8) [-1.16 to -0.49] | 0.90 (2.4) [0.56 to 1.23]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -1.72, 95% CI 2-sided [-2.20 to -1.25]

7. Secondary Outcome: Percentage of Participants With HbA1C < 7.0% at Week 30
Description: HbA1C is blood marker used to report average blood glucose levels over a prolonged periods of time and is reported as a percentage (%).
Time Frame: Week 30
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Sitagliptin/Metformin | Glimepiride
Number analyzed (Participants) | 138 | 137
Percentage of Participants | 81.2 | 40.1
Statistical Analysis 1: Comparison: Sitagliptin/Metformin vs Glimepiride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in percent = 41.01, 95% CI 2-sided [30.0 to 51.0]

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Description: The APaT Population includes all randomized participants who received at least 1 dose of study medication.
Arm/Group | Sitagliptin/Metformin | Glimepiride
Serious Adverse Events (participants affected / at risk) | 8/146 | 9/144
Other Adverse Events (participants affected / at risk) | 62/146 | 54/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Metformin (N=146) | Glimepiride (N=144)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 1 (1) | 0 (0)
INFECTIVE SPONDYLITIS (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin/Metformin (N=146) | Glimepiride (N=144)
DIARRHOEA (Gastrointestinal disorders) | 15 (22) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 19 (20) | 9 (10)
NAUSEA (Gastrointestinal disorders) | 10 (12) | 4 (4)
NASOPHARYNGITIS (Infections and infestations) | 13 (19) | 17 (22)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 12 (13) | 4 (4)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 8 (12) | 29 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.